CLINICAL TRIAL: NCT06964113
Title: A Multi-center, Open-Label, Single-Arm, Phase 4 Study to Evaluate the Efficacy and Safety of Filgotinib 200 mg in Korean Patients With Moderately to Severely Active Ulcerative Colitis Under Routine Clinical Practice
Brief Title: A Study of Filgotinib 200 mg in Korean Participants With Moderately to Severely Active Ulcerative Colitis Under Routine Clinical Practice
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS6034-M082-402
Record Dates: First submitted 2025-05-02; First posted 2025-05-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
Keywords: Jyseleca; Filgotinib maleate
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Filgotinib Maleate 200 milligram per day (mg/day) (Experimental)
  Interventions: Drug: Filgotinib Maleate

INTERVENTIONS:
Drug: Filgotinib Maleate — Administered as oral tablets.
  Other Names: Jyseleca

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of filgotinib in establishing clinical remission at Week 10 or 22.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants aged 19 to 64 years at the time of written consent
2. Participants must meet both of the following conditions:

   i) Diagnosed with moderately to severely active ulcerative colitis as determined by the Mayo Clinic Score with endoscopy occurring during screening; total score must be between 6 and 12, inclusive and endoscopy sub-score greater than or equal to (>=) 2 (However, if there are results of an endoscopy performed within two (2) months of the screening visit, and if NHI evaluation can be performed using the stored specimens obtained from that endoscopy, it can replace screening endoscopy.) ii) Have had an inadequate response to, lost response to, or were intolerant to either conventional therapy (corticosteroids, immunosuppressants, etc.) or a biologic agent based on the investigator's judgement at the screening visit.
3. Participant who is considered reliable by the investigator regarding provision of information, and is willing to comply with the study protocol procedures

Exclusion Criteria:

1. Participants with hypersensitivity to the active substance or to any of the excipients listed in the approved label of filgotinib
2. Participants with active infections, including serious infections (example [e.g.], sepsis) or local infections
3. Participants with active tuberculosis (TB). For participants with latent tuberculosis, domestic standard anti-tuberculosis therapy must be initiated at least 3 weeks prior to the first administration of the study drug (Visit 2, Day 1).
4. Participants with severe hepatic impairment (Child-Pugh C)
5. Participants with moderate or greater renal impairment (Creatinine Clearance [CrCl] less than (<) 60 milliliter per minute [mL/min])
6. Participants who meet any of the following laboratory values:
7. Absolute neutrophil count (ANC) less than (<) 1*10^9 cells per liter (/L)

   * Absolute lymphocyte count (ALC) <0.5*10^9 cells/L
   * Hemoglobin level <8 grams per deciliter (g/dL)
   * Hemoglobin level <8 g/dL
8. Female participants who are pregnant or breastfeeding at Visit 1. Even if a pregnancy test result at Visit 1 was negative, a separate evaluation is required at Visit 2 if the first dose of the study drug was administered more than 72 hours after the pregnancy test.
9. Female participants of childbearing potential who do not agree to use one of the following highly effective methods of contraception from 4 weeks prior to Visit 1 until 4 weeks after the last dose of study drug:

   * Complete abstinence (if this is the preferred and usual lifestyle of the participants)
   * Intrauterine device or hormone-containing intrauterine system (IUS)
   * Contraceptive implant
   * Oral contraceptives (participants must be on the same oral contraceptive at a stable dose for at least 4 weeks prior to the administration of the study drug, during the study and for 4 weeks after discontinuation of the study drug)
   * Partner has had a vasectomy and is confirmed to be azoospermia If a highly effective method of contraception is not appropriate or acceptable for the participants, the participants must agree to use a medically acceptable method of contraception, that is (i.e.), double barrier method of contraception such as latex or synthetic condom plus diaphragm or cervical/vault cap with spermicide.

   Note: All women will be considered to be of childbearing potential unless they are postmenopausal (at least 12 consecutive months of amenorrhea with no other known or suspected cause) or surgically sterile (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all surgically performed, at least 1 month prior to the administration of the study drug).
10. Participants with hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption
11. Participants with a history of prior treatment with Janus kinase (JAK) inhibitor
12. Participants currently participating in other clinical study or participants who used other investigational product/medical device within 4 weeks of the screening visit
13. Participants deemed inappropriate to participate in this study at the investigator's discretion.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 10 or 22 | At Week 10 or 22

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Weeks 10, 22 and 58 | At Weeks 10, 22 and 58
Percentage of Clinical Responders at Week 10 and 22 | At Week 10 and 22
Percentage of Participants Achieving Sustained Clinical Remission at Week 58 | At Week 58
Percentage of Participants Achieving Mayo Clinic Score (MCS) Remission at Weeks 10, 22, and 58 | At Weeks 10, 22, and 58
  MCS remission is defined as a MCS of 2 or less and no single sub-score higher than 1 at each time of evaluation.
Percentage of Participants Achieving Endoscopic Subscore of 0 at Weeks 10, 22, and 58 | At Weeks 10, 22, and 58
Percentage of Participants Achieving Nancy Histologic Index (NHI) Histologic Remission at Weeks 10, 22, and 58 | At Weeks 10, 22, and 58
Percentage of Participants Achieving MCS Remission (Alternative Definition) at Weeks 10, 22, and 58 | At Weeks 10, 22, and 58
  MCS remission (alternative definition) is defined as rectal bleeding (RB), stool frequency (SF), and physician's global assessment (PGA) sub-scores of 0 and an endoscopic sub-score of 0 or 1 (overall MCS of less than or equal to [<=1]) at each time of evaluation.
Percentage of Participants Achieving 6-month Corticosteroid-free Clinical Remission at Week 58 | At Week 58
Number of Participants With Adverse Events (AEs) | Up to 62 weeks
Number of Participants With Clinically Significant Abnormal Laboratory Tests | Up to 62 weeks
Number of Participants With Clinically Significant Abnormal Vital Signs | Up to 62 weeks
Number of Participants With Clinically Significant Abnormal Weight | Up to 62 weeks
Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Measurements | Up to 62 weeks
Duration of Filgotinib Exposure | Up to 58 weeks
Percentage of Participants Who Complied to Treatment | Up to 58 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- South Korea (18):
  - Eisai Site #13, Busan
  - Eisai Site #15, Busan
  - Eisai Site #8, Busan
  - Eisai Site #6, Daegu
  - Eisai Site #2, Daejeon
  - Eisai Site #16, Gyeonggi-do
  - Eisai Site #18, Jungnam
  - Eisai Site #7, Jungnam
  - Eisai Site #10, Seoul
  - Eisai Site #12, Seoul
  - Eisai Site #14, Seoul
  - Eisai Site #19, Seoul
  - Eisai Site #1, Seoul
  - Eisai Site #3, Seoul
  - Eisai Site #5, Seoul
  - Eisai Site #9, Seoul
  - Eisai Site #4, Suwon
  - Eisai Site #11, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.